CLINICAL TRIAL: NCT02332057
Title: Diclofenac Plus Lidocaine Gel for Pain Relief During Intrauterine Device (IUD) Insertion. A Randomized Double Blinded Placebo-controlled Study
Brief Title: Diclofenac Plus Lidocaine Gel for Pain Relief During Intrauterine Device Insertion(IUD).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Usama M Fouda, M.D, PhD, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Diclofenac/lidocaine/IUD
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Pain
Keywords: IUD,Diclofenac , Lidocaine
MeSH Terms: conditions — Pain | interventions — Diclofenac; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diclofenac plus lidocaine (Active Comparator): Diclofenac(100 mg) is administered 1 hour before IUD insertion and lidocaine gel is placed on cervix three minutes before IUD insertion
  Interventions: Drug: Diclofenac plus lidocaine
- Placebo (Placebo Comparator): Placebo tablets is administered 1 hour before IUD insertion and placebo gel is placed on cervix three minutes before IUD insertion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac plus lidocaine — The study nurse will instruct the patients to swallow diclofenac tablets (100 mg) 1 hour before IUD insertion. Three millilitres of the lidocaine gel will be placed on the anterior lip of the cervix . A cotton swab socked in 3 ml of the lidocaine gel will be introduced in the cervical canal till the level of internal os. The cotton swab will be left in place for three minutes. The IUD will be inserted by experienced gynecologists according to the recommendations of manufacture.
  Arms: Diclofenac plus lidocaine
Drug: Placebo — The study nurse will instruct the patients to swallow placebo tablets 1 hour before IUD insertion. Three millilitres of the placebo gel will be placed on the anterior lip of the cervix . A cotton swab socked in 3 ml of the placebo gel will be introduced in the cervical canal till the level of internal os. The cotton swab will be left in place for three minutes. The IUD will be inserted by experienced gynecologists according to the recommendations of manufacture.
  Arms: Placebo

SUMMARY:
The aim of this study is to determine the effectiveness of a combination of diclofenac and lidocaine gel in reducing pain during IUD insertion.

DETAILED DESCRIPTION:
Various studies evaluating the use of local anesthetics or misoprostol prior to IUD insertion have mixed results.We think that the combination of diclofenac and lidocaine gel could be more successful in relieving pain during IUD insertion than single therapy.The aim of this study is to determine the effectiveness of a combination of diclofenac and lidocaine gel in reducing pain during IUD insertion.

ELIGIBILITY:
Inclusion Criteria:

* Patients of reproductive age requesting IUD for contraception

Exclusion Criteria:

* Patients with contraindications to IUD insertion ( less than 6 weeks postpartum, less than 2 weeks after abortion, uterine anomalies, fibroid distorting uterine cavity, pregnancy, pelvic inflammatory disease, cervicitis, uterine depth less than 6 cm or more than 9 cm) , previous IUD insertion, allergy to diclofenac or lidocaine, peptic ulcer , asthma, bleeding disorders, cardiac, liver or kidney diseases.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Intensity of pain | Pain intensity will be assessed by visual analogue scale during the procedure [an expected average of 3 minutes]

SECONDARY OUTCOMES:
Adverse effects of diclofenac and lidocaine | Within 24 hours after IUD insertion

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, M.D,PhD, Study Chair — Cairo University
Locations (1):
- Obstetrics and Gynecology Department,Cairo university, Cairo, Egypt

REFERENCES:
- [Background] McNicholas CP, Madden T, Zhao Q, Secura G, Allsworth JE, Peipert JF. Cervical lidocaine for IUD insertional pain: a randomized controlled trial. Am J Obstet Gynecol. 2012 Nov;207(5):384.e1-6. doi: 10.1016/j.ajog.2012.09.018. Epub 2012 Sep 20. PMID 23107081
- [Derived] Fouda UM, Salah Eldin NM, Elsetohy KA, Tolba HA, Shaban MM, Sobh SM. Diclofenac plus lidocaine gel for pain relief during intrauterine device insertion. A randomized, double-blinded, placebo-controlled study. Contraception. 2016 Jun;93(6):513-8. doi: 10.1016/j.contraception.2016.02.001. Epub 2016 Feb 4. PMID 26852833